CLINICAL TRIAL: NCT01314209
Title: Dexmedetomidine Pharmacokinetics During Continuous Venovenous Hemodialysis in Critically Ill Patients
Brief Title: Dexmedetomidine Pharmacokinetics During Continuous Renal Replacement Therapy (CRRT)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Kirsi-Maija Kaukonen, Division of Anaesthesia and Intensive Care Medicine, Department of Surgery, Helsinki University Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11102010
Record Dates: First submitted 2011-03-08; First posted 2011-03-14 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2011-03

CONDITIONS: Acute Kidney Injury
Keywords: dexmedetomidine; pharmacokinetics; critical illness; continuous renal replacement therapy
MeSH Terms: conditions — Acute Kidney Injury; Critical Illness | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dexmedetomidine (Experimental)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine 0.7 microg/kg/h 12-hour intravenous infusion

SUMMARY:
The purpose of this study is to determine dexmedetomidine pharmacokinetics during continuous renal replacement therapy on critically ill patients.

DETAILED DESCRIPTION:
Dexmedetomidine is a selective alpha-2-adrenergic agonist with sedative properties indicated for sedation of patients in the intensive care setting. ICU patients with acute kidney injury requiring renal replacement therapies frequently have changes in volume status causing alterations in drug pharmacokinetics. Although dexmedetomidine pharmacokinetics have been studied earlier on ICU patients, there is no information on its pharmacokinetics in critically ill patients needing continuous renal replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Clinical need for sedation
* Acute kidney injury requiring renal replacement therapy (according to ICUs standard operating procedures)

Exclusion Criteria:

* Severe bradycardia (HR < 50/min)
* AV conduction block II-III (unless pacemaker installed)
* Severe hepatic impairment (bilirubin > 101 umol/l)
* Pregnancy or lactation
* Age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2011-03; Primary Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Dexmedetomidine clearance by continuous venovenous hemodialysis | 10 hours from the start of the dexmedetomidine infusion

CONTACTS AND LOCATIONS:
Overall Officials: Kirsi-Maija Kaukonen, MD, PhD, Principal Investigator — Division of Anaesthesia and Intensive Care Medicine, Department of Surgery, HUCH
Locations (1):
- Meilahti Hospital, Division of Anaesthesia and Intensive Care Medicine, Department of Surgery, Helsinki University Central Hospital, Helsinki, Finland